CLINICAL TRIAL: NCT05709821
Title: IMPORT-201: A Phase 1 First-in-Human Dose Finding/Randomized Phase 2 Study of IMM60 and Pembrolizumab for Advanced Melanoma and Metastatic NSCLC
Brief Title: IMM60 and Pembrolizumab in Melanoma and NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Prioritization of other pipeline assets. No safety or efficacy issues were observed.
Sponsor: iOx Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Portage Biotech (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPORT-201; KEYNOTE-E69 (Other: Merck Sharp & Dohme LLC); 2022-003310-36 (EudraCT Number)
Record Dates: First submitted 2023-01-06; First posted 2023-02-02 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; Melanoma
Keywords: Invariant natural killer T cells (iNKT); Programmed Cell Death-1 (PD1, PD-1)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 IMM60 dose escalation safety arm (Experimental): 3 dose levels of IMM60 will be assessed (1, 3, 9 and 36 mg/m^2 administered IV every 3 weeks for up to 6 cycles)
  Interventions: Drug: IMM60
- Phase 1 IMM60 + pembrolizumab combination safety arm (Experimental): Pembrolizumab 200 mg IV every 3 weeks for up to 35 cycles will be administered in combination with IMM60 IV every 3 weeks for up to 6 cycles. The IMM60 dose will be determined based on the results of the IMM60 dose escalation safety cohort.
  Interventions: Drug: IMM60; Drug: Pembrolizumab
- Phase 2 PD-L1 ≥50% NSCLC Cohort 1 (Randomized, IMM60 + pembrolizumab) (Experimental): Pembrolizumab 200 mg IV every 3 weeks for up to 35 cycles will be administered in combination with IMM60 IV every 3 weeks for up to 6 cycles. The IMM60 dose will be determined based on the results of the Phase 1 dose escalation safety cohorts.
  Interventions: Drug: IMM60; Drug: Pembrolizumab
- Phase 2 PD-L1 ≥50% NSCLC Cohort 1 (Randomized, pembrolizumab monotherapy) (Active Comparator): Pembrolizumab 200 mg IV every 3 weeks for up to 35 cycles.
  Interventions: Drug: Pembrolizumab
- Phase 2 PD-L1 <1% NSCLC Cohort 2 (Experimental): Participants will be treated with one cycle of IMM60 with a tumor biopsy before and after, to determine any changes in PD-L1 expression. After this one cycle, the participants will receive the combination of IMM60 IV for up to 6 total cycles + pembrolizumab 200 mg every 3 weeks administered IV. The IMM60 dose will be determined based on the results of the Phase 1 dose escalation cohorts.
  Interventions: Drug: IMM60; Drug: Pembrolizumab
- Melanoma Cohort (Experimental): IMM60 IV every 3 weeks for up to 6 cycles. The IMM60 dose will be determined based on the results of the Phase 1 dose escalation cohorts.
  Interventions: Drug: IMM60

INTERVENTIONS:
Drug: IMM60 — IMM60, every 3 weeks for up to 6 cycles, intravenous (IV) infusion
  Other Names: PORT-2
  Arms: Melanoma Cohort; Phase 1 IMM60 + pembrolizumab combination safety arm; Phase 1 IMM60 dose escalation safety arm; Phase 2 PD-L1 <1% NSCLC Cohort 2; Phase 2 PD-L1 ≥50% NSCLC Cohort 1 (Randomized, IMM60 + pembrolizumab)
Drug: Pembrolizumab — Pembrolizumab, 200 mg, every 3 weeks for up to 35 cycles or approximately 2 years, intravenous (IV) infusion
  Other Names: KEYTRUDA®
  Arms: Phase 1 IMM60 + pembrolizumab combination safety arm; Phase 2 PD-L1 <1% NSCLC Cohort 2; Phase 2 PD-L1 ≥50% NSCLC Cohort 1 (Randomized, IMM60 + pembrolizumab); Phase 2 PD-L1 ≥50% NSCLC Cohort 1 (Randomized, pembrolizumab monotherapy)

SUMMARY:
The goal of this clinical trial is to learn about IMM60 with or without pembrolizumab in participants with advanced melanoma or non-small cell lung cancer. There are two phases:

* Phase 1: This phase is designed to learn about the safety of IMM60 with or without pembrolizumab and to find a safe dose to test in Phase 2.
* Phase 2: This phase is designed to learn whether IMM60 + pembrolizumab improves progression-free survival at 12 months compared to pembrolizumab alone in participants with non-small cell lung cancer.

DETAILED DESCRIPTION:
This exploratory phase 1/phase 2 study is designed to establish a recommended phase 2 dose of IMM60 and provide preliminary estimates of safety and efficacy of IMM60 alone and in combination with pembrolizumab in participants with NSCLC and melanoma. In phase 1, initial safety will be assessed in a multiple dose escalation cohort for IMM60 alone, then for the IMM60 + pembrolizumab combination. Phase 2 of the study will recruit PD-1 pretreated melanoma participants and randomize PD-L1 > 50% total NSCLC participants 2:1 to IMM60 + pembrolizumab vs pembrolizumab alone. There is an additional cohort of PD-L1 < 1% NSCLC participants.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score 0 to 1
* Adequate organ function
* At least 1 lesion, not previously irradiated, that can be accurately measured on CT or MRI as defined by RECIST 1.1 criteria
* NSCLC cohorts: Histologically confirmed diagnosis of stage IV NSCLC
* NSCLC cohorts: Patients with adenocarcinoma histology must not have sensitizing epidermal growth factor receptor (EGFR) or ROS proto-oncogene 1 (ROS1) mutations or anaplastic lymphoma kinase (ALK) translocations
* NSCLC cohorts: Participants in NSCLC arms must have a PD-L1 assessment (PD-L1 immuno-histochemistry (IHC) 22C3 pharmDx)
* Melanoma cohorts: Unresectable stage III or IV, histologically confirmed diagnosis of cutaneous or unknown primary melanoma
* Melanoma cohorts: B-type Raf proto-oncogene (BRAF) mutation status available
* Male participants: Participant must agree to use contraception and refrain from sperm donation during the treatment period and for at least 120 days after the last dose of study intervention
* Female participants: Participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  1. Not a woman of childbearing potential (WOCBP)
  2. A WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 6 months after the last dose of study intervention

Exclusion Criteria:

* Has the following cardiac conditions:

  1. Corrected QT interval (QTc) > 450 ms
  2. Uncontrolled hypertension with blood pressure (BP) > 160/100 despite treatment
  3. Class II or greater heart failure as defined by the New York Heart Association
  4. Myocardial infarction within 6 months or angina requiring nitrate therapy more than once a week
* Another active malignancy within the past 2 years (Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder, or carcinoma in situ [e.g., breast carcinoma, cervical cancer in situ] that have undergone potentially curative therapy are not excluded. Also, prostate, breast, and neuroendocrine tumors that are stable on hormonal treatment for a period of 1 year or more without the need to adjust dose are not excluded.)
* Has had an allogeneic tissue/solid organ transplant
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Participants with an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids (in dosing exceeding 10 mg daily of prednisone equivalent) or immunosuppressive agents.
* Participants who are known to be serologically positive for Hepatitis B, Hepatitis C, or human immunodeficiency virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Phase 1 Co-Primary Objective - Identify Maximum Tolerated Dose (MTD) | Assessed at the end of Cycle 1 for each patient (each Cycle is 28 days)
  To confirm the maximum tolerated dose (MTD) of IMM60 alone and in combination with pembrolizumab, defined as the highest dose level at which <2 out of 6 participants experience a dose-limiting toxicity
Phase 1 Co-Primary Objective - Safety | Through Phase 1 completion, an average of 1 year
  To characterize the safety of IMM60 alone and in combination with pembrolizumab, as assessed by the frequency of Grade 3 or higher treatment-related adverse events
Phase 2 Primary Objective - Progression-free Survival | 12 months after last participant enrolled
  To compare the progression-free survival (PFS) rate at 12 months in the randomized arms comparing pembrolizumab alone versus IMM60 + pembrolizumab in patients with advanced PD-L1 ≥50% NSCLC

SECONDARY OUTCOMES:
To characterize the safety of IMM60 alone or in combination with pembrolizumab | Through study completion, an average of 3 years
  Frequency and severity of treatment-related adverse events (AEs)
To determine if IMM60 can restore sensitivity in PD-1 inhibitor-resistant melanoma (phase 2) | 12 months after last participant enrolled
  Objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 in melanoma patients who have progressed on PD-1, and have added IMM60
Pharmacokinetics of IMM60 - Cmax (IMM60 arms only) | During Cycles 1 and 3 (each Cycle is 28 days)
  IMM60 maximal concentration (Cmax)
Pharmacokinetics of IMM60 - AUC (IMM60 arms only) | During Cycles 1 and 3 (each Cycle is 28 days)
  IMM60 area under the curve (AUC)
Objective Response Rate (ORR) | 12 months after last participant enrolled
  ORR is to be reported as the proportion of patients who have a Complete Response or Partial Response per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
To determine if IMM60 can sensitize patients with programmed death-ligand 1 (PD-L1) <1% NSCLC to PD-1 inhibition | 12 months after last participant enrolled
  Objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 in PDL1 <1% NSCLC patients who receive IMM60 + pembrolizumab
To assess the ability of IMM60 to convert PD-L1 negative patients to PD-L1 positive | 12 months after last participant enrolled
  Percent of PD-L1 negative (<1%) NSCLC tumors that increase PD-L1 gene expression following treatment with IMM60

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Dana-Farber Cancer Institute - Medicine, Boston, Massachusetts
  - Henry Ford Hospital - Internal Medicine, Detroit, Michigan
  - Rutgers, The State University of New Jersey - Robert Wood Johnson Medical School - The Cancer Institute of New Jersey (CINJ), New Brunswick, New Jersey
  - Next VA, Fairfax, Virginia
- Spain (8):
  - Institut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Xeral Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen De La Macarena, Seville
  - H. Clínico de Valencia, Valencia
- Nottingham University Hospital - Oncology, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided